CLINICAL TRIAL: NCT06596057
Title: Head of Hematology，Vice President and Secretary-General of Shandong Stem Cell Society
Brief Title: Safety and Efficacy of CD19 CAR-T/CAR-NK Cells
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Linlin Cui, professor of medicine, The Second Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024CAR-T/NK B-nhl/ALL
Record Dates: First submitted 2024-08-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Safety and Efficacy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Biological: CAR-T/CAR-NK cells

INTERVENTIONS:
Biological: CAR-T/CAR-NK cells — One to two days after completion of eluvial chemotherapy, CAR-T/CAR-NK cells were transfused in subjects assessed by the investigators as eligible for infusion. The CAR-T/CAR-NK dose is calculated according to the patient's body weight, and the total number of cells transfused is about 1-2x106 /kg. Single intravenous infusion

SUMMARY:
To investigate the safety and efficacy of CD19 CAR-T/CAR-NK cells in patients with relapsed/refractory B-cell lymphoma and acute B-lymphoblastic leukemia.

DETAILED DESCRIPTION:
Patients who met the exclusion criteria were treated with advanced FC regimen, and subjects who met the infusion criteria assessed by the investigators were given CAR-T/CAR-NK cell infusion 1 to 2 days after completion of eluvial chemotherapy. The CAR-T/CAR-NK dose is calculated according to the patient's body weight, and the total number of cells transfused is about 1-2x106 /kg. Single intravenous infusion.

The study was divided into five stages: screening period, single harvest period, pretreatment chemotherapy period, treatment period, observation and follow-up period after treatment.

For lymphoma, refer to the 2014 version of Lugano efficacy evaluation criteria

ELIGIBILITY:
Inclusion criteria 1) CD19-positive recurrent, refractory, drug-resistant B-cell lymphoma and acute B-lymphoblastic leukemia. 2) Recurrent MRD-positive refractory acute B lymphoblastic leukemia, extramedullary leukemia lesions. 3) Age over 15 and under 80. 4) KPS≥50 or ECOG score ≤2 and expected survival greater than 3 months. 5) At least 2 weeks prior to apheresis or at least 5 drug half-lives (whichever is shorter) without systemic therapy (except systemic immune checkpoint suppression or activation therapy). 6) The absolute number of neutrophils is greater than 1.5x109 /L. 7) The absolute number of platelets is greater than 50x109 /L. 8) The absolute number of lymphocytes is greater than or equal to 0.15x109 /L. 9) ALT/AST is less than 3 times the normal value. 10) Total bilirubin less than 1.5mg/dl. 11) Creatinine less than 2.5mg/dl, or creatinine clearance ≥60 mL/min/1.73 m2. 12) The ejection fraction of the heart was greater than or equal to 45%, no pericardial effusion was found without echocardiography (ECHO), and electrocardiogram (ECG) was normal. 14) Blood oxygen saturation is greater than or equal to 92% under normal conditions. 15) No central nervous system metastasis was found in patients with central nervous system leukemia and lymphoma (symptoms, signs, imaging, cerebrospinal fluid). 16) Women of childbearing age who had a negative urine pregnancy test before dosing began and agreed to take effective contraception during the trial until the last follow-up visit. 17) Volunteer to participate in this experiment and sign the informed consent.

Exclusion criteria

1. Patients with expected survival of less than 3 months.
2. Clinical findings (symptoms, signs, imaging, cerebrospinal fluid) of central nervous system leukemia.
3. Patients with hyperleukocytoemia (white blood cell count ≥50 x109 /L) or patients whose disease is progressing rapidly at the time of enrollment, as determined by the investigator, to be unable to ensure the completion of a full treatment cycle.
4. Patients with skin cancer other than melanoma or other primary tumors (such as cervical cancer, bladder cancer, breast cancer) (unless cured for more than 3 years).
5. Patients with infections including fungal, bacterial, viral or other uncontrolled infections or those requiring level 4 isolation.
6. Patients who test positive for HIV, HBV, HCV.
7. Patients with central nervous system diseases including stroke, epilepsy, dementia or autoimmune central nervous system diseases.
8. Myocardial infection, cardiac angiography or stenting, active angina pectoris or other obvious clinical symptoms, or cardiac asthma or cardiovascular lymphocyte infiltration in the 12 months prior to enrollment.
9. Those who are receiving anticoagulation therapy or have severe coagulation dysfunction.
10. According to the investigator's judgment, the drug treatment the patient is receiving will affect the safety and efficacy study of this project.
11. Patients with allergy or history of allergy to the biologics used in this project.
12. Pregnant or lactating women.
13. Systematic use of systemic or systemic steroid drugs within 2 weeks prior to treatment (except those who have recently or currently used inhaled steroids).
14. The efficiency of T cell transduction by replication-deficient lentivirus is less than 30%, or the ability to expand in response to CD3 / CD28 costimulatory signals is insufficient (<5 times).
15. Those who have other uncontrolled diseases that the researchers consider unsuitable for enrollment.
16. Any situation that the investigator believes may increase the risk to the subject or interfere with the test results.
17. Patients who are also participating in other clinical studies.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
ORR | At least half a year
  With reference to iRecist1.1, the proportion of patients whose tumor volume shrank to the pre-specified value and maintained the minimum time limit.The time from randomization to tumor progression or death from any cause.
PFS | one year
  In tumor therapy, the proportion of patients whose tumor volume has shrunk to a predetermined value and can be maintained for a certain time. It includes the number of patients with complete response (CR) and partial response (PR) as a proportion of the total number of evaluable cases

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Province, Shandong, Shandong, China